CLINICAL TRIAL: NCT03799185
Title: Dyslipidemia Prevalence, Perception, Treatment, and Awareness in the Tunisian Population : The ATERA Survey
Brief Title: Dyslipidemia Prevalence, Perception, Treatment, and Awareness in the Tunisian Population
Acronym: ATERASurvey
Status: Completed | Type: Observational
Sponsor: Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose (Other)
Collaborators: Biochimie Clinique LR99ES11 (Unknown); Department of Biochemistry, La Rabta Hospital, Tunisia. (Unknown); Ministry of Health, Tunisia (Unknown); Ministry of Interior, Tunisia (Unknown); Direction des Soins de Santé de Base (Other Government); National Institute of Statistics (Unknown); National Institute of Public Health of Tunisia (Unknown); Dacima Consulting (Other)
Responsible Party: Sponsor
Other Study IDs: ID5726367
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Dyslipidemias; Atherosclerosis; Households; Survey, Family Life
Keywords: Coronary Heart Disease; Hypercholesterolemia; Triglycerides High; LDL Hyperlipoproteinemia; HDL Low; Diabetes; Cardiovascular Diseases; Hypertension; Risk Factor, Cardiovascular; Diet Habit; Smoking
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis; Coronary Disease; Hypercholesterolemia; Hypertriglyceridemia; Diabetes Mellitus; Cardiovascular Diseases; Hypertension; Feeding Behavior; Smoking

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ATERA Survey is a national cross sectional observational study, aiming to determine the prevalence of dyslipidemia and other conventional risk factors for CHD (Coronary Heart Disease), the relationship between environmental and lifestyle factors with dyslipidemia, the perception and the knowledge of cardiovascular risk factors by the population, and above all, to strengthen the national strategy for primary and secondary prevention against coronary heart disease.

DETAILED DESCRIPTION:
ATERA Survey is carried on in a random sampling including 10 000 men and women from the seven regions of Tunisia (Great Tunis, North East, North West, central East, Central West, South East and South West. The screening is being assessed using surveys covering socioeconomic, nutritional and anthropometric measures in addition to biological assessments.

The target population is being recruited by random sampling drown by the National Institute of Statistics (Tunisia). The estimated number of participants at the end of recruitment amount to 10 000. The frame sampling uses a two stage cluster sampling (district and household).

Interview with each eligible participant will be conducted mainly during assessment visit and after consenting the subject, it will be notified all the demographic, behavioral history, family history, cardiovascular risk factors and medical history. During the assessment visit, Physical examination/anthropometry data and Diet survey will be filled up by the investigator.

Data capture will be performed by the DACIMA Clinical Suite according to FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation)

ELIGIBILITY:
Inclusion Criteria:

* All subjects

Exclusion Criteria:

* Prescribed treatment for cancer
* Organ transplantation
* Known auto-immune disease
* Severe liver disease
* Chronic renal failure
* Pregnant women

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects aged between 25 and 75 years who accept to participate at the study
Sampling Method: Probability Sample
Enrollment: 13610 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of dyslipidemia | At inclusion
  Frequency of subjects with hypercholesterolemia and/or hypertriglyceridaemia

SECONDARY OUTCOMES:
Prevalence of cardiovascular associated risk factors | At inclusion
  Frequency of subjects with cardiovascular risk factors (diabetes, hypertension, obesity, gender, smoking)

OTHER OUTCOMES:
Dietary assessment | Up to 1 month
  Frequency of diet daily intake (fat, sugar, proteins, fiber)

CONTACTS AND LOCATIONS:
Overall Officials: Amani Kallel, PhD, Study Chair — Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose; Riadh Jemaa, PhD, Study Chair — Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose
Locations (1):
- ATERA : Association Tunisienne d'Etude & de Recherche sur l'Athérosclérose, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
CSR (Clinical Study Report)